CLINICAL TRIAL: NCT06130982
Title: Effects of Different Health Qigong Routines on Cervical Spondylosis Among Chinese College Students
Brief Title: Effects of Different Health Qigong Routines on CS Among Chinese College Students
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Universiti Putra Malaysia (Other)
Responsible Party: Principal Investigator, Liu Cong, Principal Investigator, Universiti Putra Malaysia
Allocation: Randomized | Model: Sequential | Masking: Triple | Purpose: Basic Science
Other Study IDs: Liu Cong
Record Dates: First submitted 2023-11-08; First posted 2023-11-14 (Actual); Last update posted 2023-11-14 (Actual); Status verified 2023-11

CONDITIONS: Neck Pain; Neck Disorder; Cervical Spondylosis
Keywords: Health Qigong; Cervical Syndrome; Curative Effect
MeSH Terms: conditions — Neck Pain; Spondylosis | interventions — Walking

STUDY DESIGN:
Intervention Model Description: In this experiment, the experimental group intervened in the content of different Health Qigong routines designed in this study. In contrast, the control group intentionally intervened in walking exercise.
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- EG1:Health Qigong·Yijinjing (Experimental): HQ·Yijinjing includes the following 10 movements:Wei Tuo Presenting the Stick1-3,Picking the star and Embracing the Moon,Hauling Nine Cattle's Tails Inversely,Pushing out the Palms Like Birds Extending the wings,Nine Ghosts Pulling Horse Blade Technique,Three Trays Falling Down,Black Dragon Streching out the Claws,Crouched Tiger,Pouncing on Its Prey,Bowing Posture,Hips Hanging.
  Interventions: Behavioral: Health Qigong·Yijinjing
- EG2:Health Qigong·Wuqinxi (Experimental): HQ·Wuqinxi includes the following 10 movements:Tiger Lifting,Tiger Pouncing,Deer Wrestling,Deer Dashing,Bear Lumbering,Bear Swaying,Monkey Hooking,Monkey Picking,Crane Stretching,Crane Flying.
  Interventions: Behavioral: Health Qigong·Wuqinxi
- EG3:Health Qigong·Baduanjin (Experimental): HQ·Baduanjin includes the following 8 movements:Supperting the Palms to the Sky to Regulate Qi of Sanjiao,Forward Lunge on the Right and Left Like Shooting an Eagle,Lifting One Arm to Regulate the Functions of Spleen and Stomach,Looking Backward to Treat Strain and Impairments,Swaying the Head and the Bottoms to Clear the Heat of Heart,Hands Grabbing Toes to Strengthen the Kidney and the Waist,Clenching Fists with Wild Eyes Glowering to Increase Strength,Raising and Lowering the Heels 7times to Alleviate Diseases.
  Interventions: Behavioral: Health Qigong·Baduanjin
- CG:Walking (Other): The control group underwent walking exercise, with a walking speed of 1.0 ± 0.2m/s based on age characteristics and human dynamic stability.
  Interventions: Behavioral: Walking

INTERVENTIONS:
Behavioral: Health Qigong·Yijinjing — 1-2weeks:learning stage, the frequency is 1 time/day, 5times/week,30 min /time,the total duration controlled within 50 minutes,and includes 4 intervention contents.Warm up activity:take a slow walk around the track and field to activate body and activate small joints (5min).Basic Skills learning of HQ·Yijinjing:breathing exercises,hand exercises,trunk exercises,step exercises,stake exercises(10min).Learning a single action of a routine (30min).Cool down (5min).3-8weeks:practice stage,the frequency and duration of intervention remain unchanged, and the intervention components still include 4 parts.Based on the first two weeks,the intervention content emphasizes more on the practice of complete routine movements, as well as learning and experience the theories and functions of movements.8-12weeks:stop intervention phase,the subjects resume their daily activities and stop intervention. After this, the final data measurement and collection are conducted again.
  Arms: EG1:Health Qigong·Yijinjing
Behavioral: Health Qigong·Wuqinxi — 1-2weeks:learning stage, the frequency is 1 time/day, 5times/week,30 min /time,the total duration controlled within 50 minutes,and includes 4 intervention contents.Warm up activity:take a slow walk around the track and field to activate body and activate small joints (5min).Basic Skills learning of HQ·Wuqinxi:breathing exercises,hand exercises,trunk exercises,step exercises,stake exercises(10min).Learning a single action of a routine (30min).Cool down (5min).3-8weeks:practice stage,the frequency and duration of intervention remain unchanged, and the intervention components still include 4 parts.Based on the first two weeks,the intervention content emphasizes more on the practice of complete routine movements, as well as learning and experience the theories and functions of movements.8-12weeks:stop intervention phase,the subjects resume their daily activities and stop intervention. After this, the final data measurement and collection are conducted again.
  Arms: EG2:Health Qigong·Wuqinxi
Behavioral: Health Qigong·Baduanjin — 1-2weeks:learning stage, the frequency is 1 time/day, 5times/week,30 min /time,the total duration controlled within 50 minutes,and includes 4 intervention contents.Warm up activity:take a slow walk around the track and field to activate body and activate small joints (5min).Basic Skills learning of HQ·Baduanjin:breathing exercises,hand exercises,trunk exercises,step exercises,stake exercises(10min).Learning a single action of a routine (30min).Cool down (5min).3-8weeks:practice stage,the frequency and duration of intervention remain unchanged, and the intervention components still include 4 parts.Based on the first two weeks,the intervention content emphasizes more on the practice of complete routine movements, as well as learning and experience the theories and functions of movements.8-12weeks:stop intervention phase,the subjects resume their daily activities and stop intervention. After this, the final data measurement and collection are conducted again.
  Arms: EG3:Health Qigong·Baduanjin
Behavioral: Walking — 1-8weeks:While the experimental group received intervention, the control group underwent walking exercise. The intervention frequency is the same as the experimental group: 1 time/day, 5times/week,30 minutes/time, the total duration controlled within 50 minutes, and includes 3 contents.Warm up activity:head movements,neck movements,shoulder movements, chest expansion exercise,waist rotation,body rotation, lunge movements,leg movements,knee joint movements,ankle movements(15 min).Walk around the track and field (30 min).Cool down (5min) 8-12weeks:stop intervention phase,the subjects resume their daily activities and stop intervention. After this, the final data measurement and collection are conducted again.
  Arms: CG:Walking

SUMMARY:
Health Qigong, originated from Chinese traditional guidance techniques, is known as China's "six major medical techniques" together with "stone breaking", "acupuncture and moxibustion", "massage", "medicine" and "walking on stilts" of traditional Chinese medicine, and has dual functions of sports and medicine. It mainly takes its own physical activities, breathing, and psychological regulation as its main form, improving the overall functional state of the human body through both internal and external cultivation, and improving the training practice method system of its own life movement. At present, it has 9 popular routines around the world, such as the famous Yi Jin Jing, Wu Qin Xi, Ba Duan Jin, and Liu Zi Jue. In the exercise therapy of cervical spondylosis, the exercise form of Health Qigong is similar to Tai Chi, and has greater advantages compared to other sports(Tai Chi, McKinsey, Cervical Spine Exercise, Resistance Exercise, etc). Previous studies have confirmed that Health Qigong·Yijinjing combined with acupuncture and moxibustion, massage and other intervention therapies can repair cervical muscle fibers, relieve pain and improve cervical function. Health Qigong·Wuqinxi combined with other intervention therapies can positively promote the pain index, cervical mobility, and other factors in middle-aged and elderly patients with cervical spondylosis.Health Qigong·Baduanjin combined with other intervention therapies can enhance the stability of the cervical spine and not only help alleviate anxiety, depression, and other adverse psychological states in patients with cervical spondylosis, It can also reduce the degree of cervical mobility limitation, thereby reducing patient pain, alleviating clinical symptoms, improving clinical intervention effectiveness, and reducing recurrence rate. However, most studies have combined exercise therapy with physical therapy, medication therapy, and other interventions therapies, especially the study of using Health Qigong as an independent exercise therapy to intervene in cervical spondylosis is even rarer. Therefore, this study selected Health Qigong·Yijinjing, Health Qigong·Wuqinxi, and Health Qigong·Baduanjin as independent exercise intervention projects to conduct intervention research on cervical spondylosis among college students, exploring the effects of these three Health Qigong routines on pain, cervical curvature, and cervical joint disorders of Chinese college students with cervical spondylosis.

DETAILED DESCRIPTION:
In the study, the experimental group conducted an 8-week intervention on the Health Qigong routine content according to the research design, as well as a 4-week follow-up observation. After screening, the subjects were randomly divided into three experimental groups and one control group. The control group of college students will receive an 8-week walking exercise,5 times a week for 30 minutes each time (a total of 50 minutes). Three experimental groups of college students will be trained according to the corresponding intervention content. EG1 is Health Qiong · Yijinjing, EG2 is Health Qiong · Wuqinxi, and EG3 is Health Qiong · Baduanjin, 5 times a week for 30 minutes each time (a total of 50 minutes). All groups of college students will undergo NDI and MPQ questionnaires, as well as measurements of cervical curvature and range of motion using X-rays and protractors, at the end of intervention in the first and eighth weeks, as well as follow-up in the twelfth week after intervention.Then, two Chinese Health Qigong level 1 social sports instructors will teach and supervise the movement standards of the experimental group. Each training session needs to strictly follow the participant's exercise mode, adhere to the exercise from low intensity to high intensity, from simple to difficult, from a single movement to the completion of the entire journey, and provide sufficient rest and Q&A time at the end of each intervention to avoid affecting the experimental level.

Content of Control Group:

Week 1-8: During the intervention period in the experimental group, after warm-up exercise, walk for 30 minutes on the track and field, and then cool down. Warming up exercise includes:head movements,neck movements,shoulder movements,chest expansion exercise,waist rotation,body rotation, lunge movements,leg movements,knee joint movements,ankle movements.

Week 9-12:Stop walking and resume daily activities. Collect data again after week 12.

Content of Experimental Group:

Week 1-2:According to the research design, college students from three experimental groups will learn warm-up activities, basic skills, and individual routine movements related to the corresponding routines. Among them, basic skills include breathing, hand type, step type, trunk, and pile skill. The routine actions of each experimental group vary depending on the intervention content.

Week 3-8:At this stage, after mastering the basic skills and movements of the intervention program, the college students in the three experimental groups, focus on practicing the complete routine movements, and during this process, focus on repeating movements related to the neck.

Week 9-12:Stop intervention and resume daily activities. Collect data again after week 12.

ELIGIBILITY:
Inclusion Criteria:

* College students aged 18-24 who experience discomfort symptoms such as neck pain and limited neck mobility;
* The X-ray shows changes in cervical curvature and is diagnosed as neck type of cervical spondylosis;
* The subjects have never sought medical attention or taken relevant medication due to cervical spondylosis;
* The subjects do not have a personal exercise plan or professional exercise background;
* The subjects are in good physical condition and possess basic athletic abilities.

Exclusion Criteria:

* If the subjects have experienced neck sprains in the past month or has experienced acute neck trauma during the experiment, which limits neck movement, it will be excluded;
* Subjects with shoulder periarthritis, rheumatic myofibrositis, neurasthenia, and other neck and shoulder pain not caused by cervical disc degeneration were excluded;
* If the subjects suffer from various congenital deformities, inflammation, tuberculosis, tumors, and other diseases of the bone itself that can cause discomfort in the neck, they are excluded;
* If the subjects are absent for more than 5 times, it will be considered as sample shedding and will be excluded.
* If the subjects fail to participate in any data collection on time, they will be excluded.

Ages: 18 Years to 24 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 80 (Estimated)
Dates: Start 2023-11-07 (Actual); Primary Completion 2024-02-07 (Estimated); Study Completion 2024-03-07 (Estimated)

PRIMARY OUTCOMES:
Effect of neck dysfunction among college students | Pretest: Before experiment; Mid-test: 8 weeks end; Post-test: 12 weeks end.
  Test by neck disability index (NDI) questionnaire , a total of 10 items were tested, including two parts: neck pain and related symptoms (intensity of pain, headache, concentration and sleep), and daily life activity ability (personal care, lifting heavy objects, reading, work, driving, and entertainment). The minimum score for each item is 0, and the maximum score is 5. The higher the score, the greater the degree of dysfunction. It can evaluate the cervical spine function impairment index, and when the result shows 0-20%, it indicates mild dysfunction; 21%-40%: indicates moderate dysfunction; 41%-60%: indicates severe functional impairment; 61% -80%: indicates extremely severe functional impairment; 81%-100%: indicates complete functional impairment or detailed examination of the subject for exaggerated symptoms.
Effect of neck pain among college students | Pretest: Before experiment; Mid-test: 8 weeks end; Post-test: 12 weeks end.
  Test by short-form of McGill pain questionnaire(SF-MPQ) ,which is derived from the McGill pain questionnaire and is used to measure the intensity and nature of pain currently experienced by participants. The lower the final evaluation score, the lower the pain intensity, and the higher the score, the higher the degree of pain. The score of SF-MPQ mainly consists of the Pain Rating Index (PRI), Present Pain Intensity (PPI), and the total pain score of the Visual Analog Scale(VAS). Among them, the evaluation of PRI consists of 15 descriptors (11 sensory; 4 affective), which are rated on an intensity scale as 0=none, 1=mild, 2=moderate or 3=distressing. The intensity evaluation of PPI is represented by 0-5, where 0=no pain, 1=mild, 2=discomforting, 3=horrible, 4=severe, and 5=excruciating.The final evaluation method of VAS is to use a digital scale with a length of approximately 10cm and labeled 0-10, 0 represents painless and 10 represents the most severe pain.
Effect of cervical curvature among college students | Pretest: Before experiment; Mid-test: 8 weeks end; Post-test: 12 weeks end.
  X-ray medical imaging examination is performed on the cervical spine of the subjects using cervical anteroposterior and lateral positions to observe changes in the physiological curvature and intervertebral space of the subjects' cervical spine. After obtaining medical imaging results, the Borden method is used to measure the physiological curvature depth (arc chord distance) of the cervical spine and observe the changes in cervical curvature of college students with cervical spondylosis.
Effect of cervical range of motion among college students | Pretest: Before experiment; Mid-test: 8 weeks end; Post-test: 12 weeks end.
  Measure the range of motion of the cervical spine using a support arm protractor.Cervical Range of Motion (CROM) is an important indicator for quantifying cervical function and evaluating the degree of cervical diseases, injuries, and rehabilitation. It mainly includes the measurement of the six cervical motion directions:cervical extension(0°~45°),cervical flexion(0°~45°),left and right cervical lateral flexion(0°~45°),left and right cervical rotation(0°~60°).Through objective measurement methods, record and analyze the cervical spine mobility, and summarize the impact of Health Qigong before and after intervention on the cervical spine mobility of college students with cervical spondylosis.

SECONDARY OUTCOMES:
Comprehensive efficacy evaluation after intervention | First test: 8 weeks end, calculate effective rate; Second test: 12 weeks end, calculate the recurrence rate.
  The effectiveness and persistence of Health Qigong intervention in cervical spondylosis can be tested through curative effect.According to the evaluation criteria for the efficacy of cervical spondylosis in the "Chinese Medicine Waiting Treatment Standards" issued in 1994, it is divided into three levels:cure,improvement and ineffectiveness.According to the standards and main measurement results, after the intervention in the eighth week,based on the main measurement results, the effective rate of the intervention is calculated as follows: (number of cured cases+number of improvement cases/total number of cases) *100%. Then, after the eighth week of intervention, all subjects resume their daily activities, and based on the results of the last follow-up measurement in week 12, the recurrence rate is calculated as follows: (Number of recurrence cases/total number of cases) *100%.

CONTACTS AND LOCATIONS:
Overall Officials: Cong Liu, Phd, Principal Investigator — University Putra Malaysia
Locations (1):
- Sichuan Nursing Vocational College, Chengdu, Sichuan, China

IPD SHARING:
Plan to Share IPD: No
Since this is my doctoral thesis experiment, I won't share it until l graduate.

REFERENCES:
- [Background] Zhang YP, Hu RX, Han M, Lai BY, Liang SB, Chen BJ, Robinson N, Chen K, Liu JP. Evidence Base of Clinical Studies on Qi Gong: A Bibliometric Analysis. Complement Ther Med. 2020 May;50:102392. doi: 10.1016/j.ctim.2020.102392. Epub 2020 Apr 6. PMID 32444061
- [Background] Chen X, Cui J, Li R, Norton R, Park J, Kong J, Yeung A. Dao Yin (a.k.a. Qigong): Origin, Development, Potential Mechanisms, and Clinical Applications. Evid Based Complement Alternat Med. 2019 Oct 21;2019:3705120. doi: 10.1155/2019/3705120. eCollection 2019. PMID 31772593
- [Background] Zou L, Zhong C, Xu X, Liu F, Wang C, Shi B. Effect of Baduanjin exercise on cervical spondylosis: A protocol for the systematic review of randomized controlled trials. Medicine (Baltimore). 2021 Mar 26;100(12):e24813. doi: 10.1097/MD.0000000000024813. PMID 33761641
- [Background] Dai W, Wang X, Xie R, Zhuang M, Chang X, Yang G, Yu J, Zhu L. Baduanjin exercise for cervical spondylotic radiculopathy: A protocol for systematic review and meta-analysis. Medicine (Baltimore). 2020 May;99(18):e0037s. doi: 10.1097/MD.0000000000020037. PMID 32358384
- [Background] Liu Z, Hu H, Wen X, Liu X, Xu X, Wang Z, Li L, Liu H. Baduanjin improves neck pain and functional movement in middle-aged and elderly people: A systematic review and meta-analysis of randomized controlled trials. Front Med (Lausanne). 2023 Jan 10;9:920102. doi: 10.3389/fmed.2022.920102. eCollection 2022. PMID 36703891
- [Background] Xu Z, Chen Y, Feng L, Lu Q. A Natural-Position X-Ray for Evaluating Cervical Vertebra Physiology Curvature Before and After Conservative Treatment. Med Sci Monit. 2023 May 18;29:e939480. doi: 10.12659/MSM.939480. PMID 37246624
- [Background] Vernon H, Mior S. The Neck Disability Index: a study of reliability and validity. J Manipulative Physiol Ther. 1991 Sep;14(7):409-15. PMID 1834753
- [Background] Melzack R. The short-form McGill Pain Questionnaire. Pain. 1987 Aug;30(2):191-197. doi: 10.1016/0304-3959(87)91074-8. PMID 3670870
- See also: This article is from National Library of Medicine. — http://pubmed.ncbi.nlm.nih.gov/32444061/
- See also: This article is from National Library of Medicine. — http://pubmed.ncbi.nlm.nih.gov/31772593/
- See also: This article is from National Library of Medicine. — http://pubmed.ncbi.nlm.nih.gov/33761641/
- See also: This article is from National Library of Medicine. — http://pubmed.ncbi.nlm.nih.gov/32358384/
- See also: This article is from National Library of Medicine. — http://pubmed.ncbi.nlm.nih.gov/36703891/
- See also: This article is from National Library of Medicine. — http://pubmed.ncbi.nlm.nih.gov/37246624/
- See also: This article is from National Library of Medicine. — http://pubmed.ncbi.nlm.nih.gov/1834753/
- See also: This article is from National Library of Medicine. — http://pubmed.ncbi.nlm.nih.gov/3670870/